CLINICAL TRIAL: NCT04346550
Title: Comparison of Morbidity After Laparoscopic Cholecystectomy for Acutely Inflamed Gall Bladder With and Without Drain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa International Hospital (Other)
Responsible Party: Principal Investigator, Dr. Hira Saleem, Post Graduate Resident, Principal Investigator., Shifa International Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sheikh
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Acute Cholecystitis; Pain; Morbidity, Multiple; Surgery; Drain Site Complication
Keywords: pain; Hospital stay; Drain insertion; Laparoscopic cholecystectomy; Acutely inflammed gall bladder
MeSH Terms: conditions — Cholecystitis, Acute; Pain

STUDY DESIGN:
Intervention Model Description: The study objective is to compare the frequency of pain and mean hospital stay in patients with and without drain insertion, following laparoscopic cholecystectomy for acutely inflamed gallbladder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drain Group (Active Comparator): Suction drain was placed in sub hepatic region through 5 mm lateral trocar site.
  Interventions: Other: Suction drain
- Without Drain Group (No Intervention): No drain was placed

INTERVENTIONS:
Other: Suction drain — Post operatively, in both arms including drain group and no drain group, parameters of pain was assessed by visual analog scale (VAS) from 0 (no pain) to 10 (worst pain), assessed at 1st postoperative day by the duty doctor or the nurse. VAS > 3 was considered as post surgical pain. The total number of hospital stay was noted from the day of operation till the day of discharge and discharge criteria was taken as a patient having pain as per VAS<3, no fever and tolerating oral intake
  Arms: Drain Group

SUMMARY:
The purpose of this study was to compare the frequency of pain and mean hospital stay in patients with and without drain insertion, following laparoscopic cholecystectomy for acutely inflamed gallbladder.

DETAILED DESCRIPTION:
Most hospitals in Pakistan still do not have a policy of early laparoscopic cholecystectomy in acutely inflamed gallbladder, partly because of feared higher conversion rates to open procedure and presumed increased risk of complications. There are fewer local studies to elaborate the role of drain after laparoscopic cholecystectomy for acutely inflamed gallbladder. This study was conducted to analyze the role of routine use of drains after laparoscopic cholecystectomy for acutely inflamed gallbladder. Does it offer any advantage in detecting bile leak or bleeding. Also to prove that placing drains prolongs the hospital stay and increases postoperative pain in comparison to patients in whom drain is not placed.

After being informed about the study and the potential risks, all patients giving written informed consent, underwent laparoscopic cholecystectomy using conventional 4 port method. Patients were divided in two groups by lottery method. Group A - no drain group and Group B - drain group. Post operatively parameters of pain and total hospital stay were assessed and analysed.

ELIGIBILITY:
Inclusion Criteria:

* All the patients of either sex with ages between 20 - 80 years, diagnosed with acutely inflamed gallbladder, undergoing laparoscopic cholecystectomy were included in the study

Exclusion Criteria:

* All patients having concurrent operations on other organs, or with history of previous upper abdominal surgery, or with immunodeficiency states because of liver or renal transplantation or already diagnosed with HIV infection, or surgeries requiring open conversions, or surgeries in which there was hollow visceral organ injury, or patient requiring common bile duct (CBD) exploration or patients having any bleeding disorder, or surgeries where there is doubt of cystic duct stump or CBD injury, were excluded from the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 1st post operative day
  Pain was assessed by VISUAL ANALOGUE SCALE (VAS) from 0 to 10, taking 0 SCORE FOR NO PAIN AND MAXIMUM 10 SCORE FOR WORST PAIN, assessed at 1st postoperative day by the duty doctor or the nurse. VAS > 3 was considered as post surgical pain.
Mean Hospital stay | 1st to 5th post operative day
  Number of days from the day of operation till the day of discharge and discharge criteria was taken as a patient having pain as per VISUAL ANALOGUE SCALE <3 (0 SCORE FOR NO PAIN AND MAXIMUM 10 SCORE FOR WORST PAIN), no fever and tolerating oral intake.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Saleem, FCPS Surgery, Principal Investigator — Shifa International Hospital
Locations (1):
- Shifa International Hospital, Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No